CLINICAL TRIAL: NCT00002065
Title: Depot Disulfiram for AIDS and ARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Vincent's Medical Center (Unknown)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 024A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-11

CONDITIONS: HIV Infections
Keywords: Delayed-Action Preparations; Disulfiram; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Disulfiram

INTERVENTIONS:
Drug: Disulfiram

SUMMARY:
To assess the safety and efficacy of depot disulfiram as a new treatment for AIDS and AIDS related complex.

ELIGIBILITY:
Inclusion Criteria

Patients must have a positive diagnosis of AIDS or AIDS related complex (ARC) according to the CDC criteria.

* Also patient must be:
* Able to understand the study.
* Strongly motivated to participate in the study, and willing to comply with all the conditions specified in the informed consent forms.
* Ambulatory and able to maintain an independent life outside the hospital.
* Free of clinically significant organic disease affecting neurologic, hepatic, renal, and clinical status.

Patients must be free of clinically significant organic disease affecting neurologic, hepatic, renal, and clinical status.

Patients must be free of clinically significant organic disease affecting neurologic, hepatic, renal, and clinical status.

History of alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Vincent's Med Ctr, Staten Island, New York, United States